CLINICAL TRIAL: NCT05269992
Title: Tolerance, Compliance and Acceptability to a New Nutritional Feed Comprising Real Food Ingredients
Brief Title: Childrens Real Food Tolerance Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NN001
Record Dates: First submitted 2022-02-16; First posted 2022-03-08 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Malnutrition, Child
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Real food products (Experimental): The study products are 1) a 1kcal/ml enteral tube feed provided as a 500ml ready to use enteral tube feed; 2) a 1.5kcal/ml enteral tube feed provided as a 500ml ready to use enteral tube feed, and 3) a 1.5kcal/ml oral nutritional supplement provided in a 200ml ready to drink format. This study is a prospective, longitudinal, 28-day intervention study with a 1-day baseline period aiming to recruit 60 in paediatric patients. During the intervention period, patients will receive one of the three study products (or more if deemed appropriate) for 28 days as a sole source of nutrition or alongside any additional routine nutritional management as required. As such, randomisation was not deemed suitable for this study. The appropriate study product and volume prescribed will be recommended by the investigating dietitian/nurse and agreed with the patient/parent/carer based on their clinical and nutritional requirements.
  Interventions: Other: Real food products

INTERVENTIONS:
Other: Real food products — As per arm/group descriptions.

SUMMARY:
A prospective, longitudinal, 28-day intervention study evaluating the tolerance, compliance, acceptability and safety to two new enteral tube feed and one new oral nutritional supplement based on real food ingredients (1kcal/ml and 1.5kcal/ml enteral tube feeds and a 1.5kcal/ml oral nutritional supplement).

DETAILED DESCRIPTION:
Nutritional feeds in the form of either enteral tube feeds or oral nutritional supplements are commonly used to meet the entire or partial nutritional requirements of children who demonstrate faltering growth or other medical conditions where they cannot meet their nutritional requirements sufficiently either orally or with food alone. Prescribable commercially available enteral tube feeds and oral nutritional supplements are recommended for all patient groups by the National Institute for Clinical Excellence (NICE) and other professional bodies and are based on food ingredients such as milk powder, vegetable oils and vitamin/mineral mixes however, they are processed to some degree to ensure stability, sterility and standardised nutritional content.

In recent years some patient groups have begun to administer homemade blended foods via their feeding tubes, instead of using prescribable commercially available feeds, which is especially prevalent among paediatric patients. Although recognition of this practice from professional bodies is low, anecdotal evidence does show some benefits. Nonetheless, there are concerns with this practice including compromised nutritional consistency, microbiological safety and enteral pump and tube integrity. This presents a problem for some parents who wish to provide their child with a source of nutritional support based on real food without posing any additional risks. Nutricia has recognised the changing needs of these paediatric patients and has therefore extended its existing range of paediatric feeds to include new formulations which include real food ingredients whilst still maintaining sterility and a stabilised nutritional content. These new formulations are designed for children with faltering growth/disease related malnutrition from 1 year old, are suitable as a sole source of nutrition and provide a sterile, standardised consistency and nutritional content.

A clinical trial is therefore required to evaluate the tolerance, compliance, acceptability and safety of three new enteral tube feed and oral nutritional supplement formulations, based on real food ingredients (1kcal/ml and 1.5kcal/ml enteral tube feeds and a 1.5kcal/ml oral nutritional supplement). Additional outcomes include nutritional intake, anthropometrics, and gastrointestinal health-related quality of life. This is a prospective, longitudinal, 28-day intervention study with a 1-day baseline period. During the intervention period, patients will receive the intervention feed(s) as a sole source of nutrition or alongside any additional routine nutritional management as required.

ELIGIBILITY:
Inclusion Criteria:

* Children from 1 year to 16 years of age.
* Requiring oral or enteral nutritional support from a whole protein 1kcal/ml or a 1.5kcal/ml enteral tube feed (via an existing enteral feeding tube) or oral nutritional supplement for at least 28 days.
* Expected to receive a minimum of 300kcal/day from the study product(s).
* Informed consent obtained from the patient/carer.

Exclusion Criteria:

* Total parenteral nutrition (100% of requirements).
* Allergy to any of the study product ingredients.
* Severe galactose (galactosaemia) or lactose intolerance.
* Severe hepatic, metabolic or renal dysfunction.
* Requirement for a fibre free feed.
* Requirement for a hydrolysed, elemental or any other specialised feed.
* On high intensity chemotherapy or radiation therapy, pancreatitis, chylothorax, or Inflammatory Bowel Disease.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal tolerance assessing abdominal discomfort, pain, nausea, reflux, regurgitation, gagging, retching, vomiting, constipation, diarrhoea, bloating and flatulence | 29 days
  Gastrointestinal tolerance will be assessed at baseline (day 1) in relation to patients' usual enteral tube feed, oral nutritional supplement or other nutritional regimen, and again at day 8, 15, 22 and 29 during the intervention using standardised questionnaires.Parents/carers will be asked to complete a gastrointestinal symptom score form on behalf of their child which will assess the incidence and severity of the following symptoms: abdominal discomfort, pain, nausea, reflux, regurgitation, gagging, retching, vomiting, constipation, diarrhoea, bloating and flatulence on a four-point scale (Absent, Mild, Moderate, Severe).

SECONDARY OUTCOMES:
Compliance | 29 days
  Compliance with the recommended intake of patients' currently prescribed enteral tube feed or oral nutritional supplement (if an existing user) will be assessed at baseline (day 1). Similarly, parents/carers will be asked to record how much study feed (ml) their child takes daily throughout the study period (days 2-29), which will be compared to the amount prescribed by the Dietitian
Functionality, perception and satisfaction with the study product | 29 days
  The acceptability of any enteral tube feeds and oral nutritional supplements used prior to study enrolment will be recorded at baseline (day 1) and consequently study products (including perceptions around enteral tube feeding and oral nutritional supplements) will be recorded at the end of week 1 and at the end of the study period (day 29) by parents/carers using standardised questionnaires. This will assess how much users agree or disagree with various statements about the feeds such as functionality (i.e. ease of use or complications), perception and satisfaction, as well as assessing changes in opinions around enteral tube feeding or oral nutritional supplements (in relation to the product taken).
Energy and protein intake | 29 days
  Energy and protein intake will be collected at baseline (day 1) and at the end of week 1 (day 8) and at the end of the study period (day 29) based on 24-hour dietary recall recorded by the Dietitian. Nutritional analysis software https://www.nutritics.com/p/home will be used to perform dietary analysis to determine energy and protein intakes.
Gastrointestinal health-related quality of life | 29 days
  Gastrointestinal health-related quality of life outcomes will be collected by parents/carers at baseline (day 1), at the end of week 1 (day 8) and end of the study period (day 29). This form will record how much users feel their enteral tube feed impacts on factors such as sleep, pain, anxiety and social functioning. Participants aged 5 years and above will also be given the opportunity (where appropriate) to give self-reported answers on a simplified version.
Height | 29 days
  Anthropometric data will be collected at baseline (day 1) and at the end of the study period (day 29), using standardised methods to assess growth. This will include weight (in kg) which will be recorded to the nearest 0.1kg. In those participants who are unable to stand on conventional weighing scales, sitting or hoist scales will be used where possible. Mid upper-arm circumference (in cm) will also be measured on a bare, relaxed arm (left) from the midpoint between the tip of the shoulder and the elbow and recorded to the nearest 0.1cm.
Weight | 29 days
  Anthropometric data will be collected at baseline (day 1) and at the end of the study period (day 29), using standardised methods to assess growth. Height (in cm) will be recorded to the nearest 0.1cm in those able to stand. Descriptive information from growth charts will also be collected to understand growth history, and growth goals will be recorded by the Dietitian.
Dietetic Goal | 29 days
  The dietetic goal of each patient will be recorded at baseline by the Dietitian and achievement of this goal (via yes/no responses) in the view of the Dietitian will be assessed at the end of the intervention (day 29).
Adverse events | 29 days
  All adverse events will be recorded throughout the study on occurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Bristol Royal Hospital for Children, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD planned. Following completion of this trial, the results may be published in conference proceedings or as a full manuscript where all data will be mean +/- SD and not individual.